CLINICAL TRIAL: NCT00703729
Title: The Effectiveness of Simultaneous Intermittent Compression and Continuous Cold Therapy on the Post-Operative Shoulder: A Randomized Controlled Trial
Brief Title: Compression and Cold Therapy on the Post-Operative Shoulder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 07-0403; 2-5-86058
Record Dates: First submitted 2008-06-19; First posted 2008-06-23 (Estimated); Results first posted 2015-09-10 (Estimated); Last update posted 2015-09-10 (Estimated); Status verified 2015-08

CONDITIONS: Postoperative Pain; Shoulder Pain
MeSH Terms: conditions — Pain, Postoperative; Shoulder Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cold Compression (CC) (Experimental): The Game Ready device provides both active, continuous cold and intermittent, pneumatic compression to the post-op shoulder. The first group will use the Game Ready™ Device (CC) for one week following surgery and will use standard ice bags wrapped to the shoulder (IW) for the remainder of the study period.
  Interventions: Device: Cold Compression (CC)
- Ice Wrap (IW) (Active Comparator): The ice bag (IW)is secured to the shoulder using an elastic wrap. The second group will use standard ice bags wrapped to the shoulder (IW) for one week following surgery and will use the Game Ready™ Device (CC) for the remainder of the study period
  Interventions: Other: Ice Wrap (IW)

INTERVENTIONS:
Device: Cold Compression (CC) — The device is applied to the shoulder within 60 minutes of arrival to the recovery room following surgery. The device will be applied at one hour intervals (60 minutes on the shoulder, 60 minutes off) during waking hours for the first 72 hours after surgery. For the remainder of the study period, therapy will be applied for one hour treatments 2-3 times a day during waking hours.
  Arms: Cold Compression (CC)
Other: Ice Wrap (IW) — The ice bag is applied to the shoulder within 60 minutes of arrival to the recovery room following surgery. The ice bag is placed on the shoulder and the elastic wrap is used to hold the bag in place. The ice will be applied at one hour intervals (60 minutes on the shoulder, 60 minutes off) during waking hours for the first 72 hours after surgery. For the remainder of the study period, therapy will be applied for one hour treatments 2-3 times a day during waking hours.
  Arms: Ice Wrap (IW)

SUMMARY:
The purpose of this study is to evaluate and compare clinical post-operative outcomes for patients using active cooling and compression device and those using ice bags and elastic wrap after acromioplasty or arthroscopic rotator cuff repair.

ELIGIBILITY:
Inclusion Criteria:

* Patient has undergone unilateral Rotator cuff repair or Acromioplasty
* Willing to sign a consent form
* Able to follow study procedures

Exclusion Criteria:

* Non-ambulatory
* Participation in concurrent investigational protocol
* Any bleeding coagulopathies
* Raynaud's disease or other vasospastic hypersensitivity or circulatory syndromes
* Hypertension (due to secondary vasoconstriction)
* Compromised local circulation (including localized compromise due to multiple surgical procedures)
* A history of vascular impairment (such as frostbite or arterial sclerosis)
* Cold allergy (cold urticaria) or prior adverse reactions to cold application
* Rheumatoid arthritis
* Local limb ischemia
* Paroxysmal cold hemoglobinuria
* Cryoglobulinemia or any disease that produces a marked cold pressor response
* Inflammatory phlebitis
* Acute inflammations of the veins (thrombophlebitis)
* Decompensated cardiac insufficiency
* Arterial dysregulation
* Erysipelas
* Deep acute venal thrombosis (phlebothrombosis)
* Carcinoma and carcinoma metastasis in the affected extremity
* Decompensated hypertonia
* Pulmonary embolisms
* Congestive heart failure
* Pulmonary edema
* Suspected deep vein thrombosis
* Acute inflammatory skin diseases
* Infection
* Venous or arterial occlusive disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2008-06; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric C McCarty, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- CU Sports Medicine, Boulder, Colorado, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cold Compression (CC) | Ice Wrap (IW)
Started | 25 | 24
Completed | 25 | 21
Not Completed | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cold Compression (CC) | Ice Wrap (IW) | Total
Number analyzed (Participants) | 25 | 24 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.4 (10.6) | 55.8 (11.2) | 55.6 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 8 | 21
  Male | 12 | 16 | 28

OUTCOME MEASURES:

1. Primary Outcome: Patient Reported Pain on Day 0
Description: Pain was measured using a visual analog scale (VAS) 10 cm in length, with "no pain" at the left side of the scale and "extreme pain" at the right side. Scores were measured to the closest millimeter for a 0-100 scale.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: Visual Analog Score (0-100)
Arm/Group | Cold Compression (CC) | Ice Wrap (IW)
Number analyzed (Participants) | 25 | 21
Visual Analog Score (0-100) | 30.2 (34.3) | 24.2 (30.0)

2. Secondary Outcome: Use of Pain Medication on Day 1
Description: Pain medication was quantified using a morphine equivalent dosage (MED) with the following scale: 1 mg of oral morphine = 1 morphine equivalent. 3 mg morphine = 3 mg hydrocodone = 2 mg oxycodone
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: Morphine Equivalent Dosage
Arm/Group | Cold Compression (CC) | Ice Wrap (IW)
Number analyzed (Participants) | 25 | 21
Morphine Equivalent Dosage | 38.6 (20.4) | 37.3 (25.2)

3. Primary Outcome: Patient Reported Pain on Day 1
Description: as for outcome 1
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: Visual Analog Score (0-100)
Arm/Group | Cold Compression (CC) | Ice Wrap (IW)
Number analyzed (Participants) | 25 | 21
Visual Analog Score (0-100) | 38.8 (24.4) | 47.4 (29.2)

4. Primary Outcome: Patient Reported Pain on Day 2
Description: as for outcome 1
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: Visual Analog Score (0-100)
Arm/Group | Cold Compression (CC) | Ice Wrap (IW)
Number analyzed (Participants) | 25 | 21
Visual Analog Score (0-100) | 34.5 (19.2) | 36.5 (29.1)

5. Primary Outcome: Patient Reported Pain on Day 3
Description: as for outcome 1
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: Visual Analog Score (0-100)
Arm/Group | Cold Compression (CC) | Ice Wrap (IW)
Number analyzed (Participants) | 25 | 21
Visual Analog Score (0-100) | 30.1 (19.5) | 33.2 (27.8)

6. Primary Outcome: Patient Reported Pain on Day 4
Description: as for outcome 1
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: Visual Analog Score (0-100)
Arm/Group | Cold Compression (CC) | Ice Wrap (IW)
Number analyzed (Participants) | 25 | 21
Visual Analog Score (0-100) | 30.6 (26.3) | 33.5 (24.5)

7. Primary Outcome: Patient Reported Pain on Day 5
Description: as for outcome 1
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: Visual Analog Score (0-100)
Arm/Group | Cold Compression (CC) | Ice Wrap (IW)
Number analyzed (Participants) | 25 | 21
Visual Analog Score (0-100) | 23.4 (19.2) | 28.0 (27.1)

8. Primary Outcome: Patient Reported Pain on Day 6
Description: as for outcome 1
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: Visual Analog Score (0-100)
Arm/Group | Cold Compression (CC) | Ice Wrap (IW)
Number analyzed (Participants) | 25 | 21
Visual Analog Score (0-100) | 27.3 (22.8) | 26.0 (26.2)

9. Primary Outcome: Patient Reported Pain on Day 7
Description: as for outcome 1
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: Visual Analog Score (0-100)
Arm/Group | Cold Compression (CC) | Ice Wrap (IW)
Number analyzed (Participants) | 25 | 21
Visual Analog Score (0-100) | 24.8 (19.9) | 23.0 (27.7)

10. Secondary Outcome: Use of Pain Medication on Day 2
Description: as for outcome 2
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: Morphine Equivalent Dosage
Arm/Group | Cold Compression (CC) | Ice Wrap (IW)
Number analyzed (Participants) | 25 | 21
Morphine Equivalent Dosage | 38.0 (28.7) | 33.2 (25.1)

11. Secondary Outcome: Use of Pain Medication on Day 3
Description: as for outcome 2
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: Morphine Equivalent Dosage
Arm/Group | Cold Compression (CC) | Ice Wrap (IW)
Number analyzed (Participants) | 25 | 21
Morphine Equivalent Dosage | 30.5 (29.8) | 28.9 (25.6)

12. Secondary Outcome: Use of Pain Medication on Day 4
Description: as for outcome 2
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: Morphine Equivalent Dosage
Arm/Group | Cold Compression (CC) | Ice Wrap (IW)
Number analyzed (Participants) | 25 | 21
Morphine Equivalent Dosage | 22.8 (29.6) | 14.3 (16.5)

13. Secondary Outcome: Use of Pain Medication on Day 5
Description: as for outcome 2
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: Morphine Equivalent Dosage
Arm/Group | Cold Compression (CC) | Ice Wrap (IW)
Number analyzed (Participants) | 25 | 21
Morphine Equivalent Dosage | 18.9 (27.9) | 11.0 (14.1)

14. Secondary Outcome: Use of Pain Medication on Day 6
Description: as for outcome 2
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: Morphine Equivalent Dosage
Arm/Group | Cold Compression (CC) | Ice Wrap (IW)
Number analyzed (Participants) | 25 | 21
Morphine Equivalent Dosage | 18.1 (26.0) | 7.7 (12.0)

15. Secondary Outcome: Use of Pain Medication on Day 7
Description: as for outcome 2
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: Morphine Equivalent Dosage
Arm/Group | Cold Compression (CC) | Ice Wrap (IW)
Number analyzed (Participants) | 25 | 21
Morphine Equivalent Dosage | 11.8 (16.7) | 6.3 (11.5)

ADVERSE EVENTS:
Arm/Group | Cold Compression (CC) | Ice Wrap (IW)
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/24
Other Adverse Events (participants affected / at risk) | 0/25 | 0/24

LIMITATIONS AND CAVEATS:
Some patients were removed from the trial due to non-compliance, most commonly for failing to complete the pain diaries.

There is also some inherent recall bias in asking a patient to fill out a diary.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No